CLINICAL TRIAL: NCT01426061
Title: Effect of Reflexology, Homeopathy and Conventional Medical Treatment in Asthma: A Randomised Controlled, Parallel Group Trial.
Brief Title: Clinical Effect of Reflexology and Homeopathy Added to Conventional Asthma Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: GCP-unit at Aarhus University Hospital, Aarhus, Denmark (Other); Danish Classical Homeopathy Society (Unknown); Danish Reflexologist Association (Other)
Responsible Party: Principal Investigator, Ayfer Topcu, M.D., University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20040206
Record Dates: First submitted 2011-08-18; First posted 2011-08-30 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Asthma
Keywords: Complementary and alternative medicine; Reflexology; Homeopathy; Asthma; Randomized controlled trial
MeSH Terms: conditions — Asthma | interventions — Musculoskeletal Manipulations; Homeopathy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Reflexology plus conventional treatment (Experimental)
  Interventions: Other: Reflexology plus conventional treatment
- Homeopathy plus conventional treatment (Experimental)
  Interventions: Other: Homeopathy plus conventional treatment
- Conventional treatment (No Intervention)
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Reflexology plus conventional treatment — Patients in the reflexology group received reflexology treatment in addition to usual care of asthma.Patients received treatments weekly for four to six weeks, followed by two treatments for one month. Treatments were then given monthly until the end of the study.
  Arms: Reflexology plus conventional treatment
Other: Homeopathy plus conventional treatment — Patients in the homeopathy group received homeopathic treatment in addition to usual care of asthma.Homeopathic treatment was decided on an individual basis by the homeopath and prescribed as an oral treatment. Patients received homeopathic product with potency between C30 (dilution by a factor 10030 =1060) and M10 (dilution by a factor 100010 =1030). The number of homeopathy sessions attended was six to twelve during one year.
  Arms: Homeopathy plus conventional treatment
Other: Conventional treatment — Patients in the conventional treatment group received usual care of asthma. This treatment was monitored and adjusted as usual by the patient's general practitioner.
  Arms: Conventional treatment

SUMMARY:
There is a lack of scientific evidence that homeopathy and reflexology is effective treatment of asthma. Systematic reviews have found that many clinical trials testing homeopathy and reflexology have major flaws, such as small number of participants, lack of control groups or inadequate allocation concealment.

The aim of the present study was to assess the effect of reflexology and individualised homeopathy as an adjuvant treatment in asthma. In order to address this issue, the investigators conducted an investigator-blinded, randomized, controlled parallel group study.

ELIGIBILITY:
Inclusion Criteria:

* Forced expiratory volume in 1 second (FEV1) ≥60% predicted
* A history of bronchial asthma for minimum 6 months prior to baseline
* An objective measure of abnormal variation in bronchial calibre(The objective measure were defined as at least one of the following)

  1. a positive bronchodilator reversibility test, defined as increase in FEV1≥10% after 400 µg inhaled salbutamol;
  2. a positive methacholine test, defined as a PD20 of <1000 μg;
  3. a positive test for exercise induced asthma defined as a fall in FEV1>15% after a standardised 6 min exercise test; and
  4. a positive peak expiratory flow (PEF) variability , defined by ≥3 days or 2 consecutive days with a differences between morning and evening PEF of >20% during a 2-week period.

Exclusion Criteria:

* Hospitalization for asthma within 3 months,
* Asthma exacerbation during the last month,
* Changes in asthma medication within 30 days of screening
* A smoking history > 10 pack-years and smoking within the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The change in the Asthma Quality of Life Questionnaire(AQLQ) | Assesment of quality of life was perfomed at baseline, at week 26 and at week 52.
  AQLQ is self-administered questionnaire which consists of 32 questions in 4 domains (symptoms, activity limitation, emotional function and environmental stimuli). Patients responded to each question on a seven point scale (7=no impairment 1=maximal impairment) and recalled their experiences during the previous 2 weeks. The overall AQLQ score was the mean of all 32 questions. A change in score of ≥0.5 indicates the minimal important difference (MID) in AQLQ.

SECONDARY OUTCOMES:
Asthma control questionnaire (ACQ) | At baseline, week 26 and week 52
EuroQol(EQ-5D) | At baseline, week 26 and week 52
Forced expiratory volume in 1 second | At baseline, week 26 and week 52
Asthma symptoms | Two weeks prior to week 2, 26 and 52.
  Daytime and nighttime symptoms were recorded in patients diaries.
Peak expiratory flow | Two weeks prior to week 2, 26 and 52.
  Morning and evening Peak expiratory flow(PEF) were performed before inhalation medication
Rescue medication usage | To weeks prior to week 2, 26 and 52
Total medication score | At baseline, at week 26 and week 52.
  Total medication score was created by combaning a score given to each prescribed controller and reliever medication.
Blood eosinophils count | At baseline, at week 26 and week 52
Exhaled nitric oxide | At baseline, at week 26 and week 52
Serum eosinophil cationic protein | At baseline, at week 26 and week 52
PD20 | At baseline, at week 26 and week 52
  The provocotive dose of Methacholine causing a 20% fall in FEV1

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dahl, MD, Principal Investigator — Department of Respiratory Diseases, University Hospital of Aarhus, DK-8000 Aarhus C
Locations (1):
- Department of Respiratory Diseases, University Hospital of Aarhus, Aarhus, Denmark

REFERENCES:
- [Background] Ng TP, Wong ML, Hong CY, Koh KT, Goh LG. The use of complementary and alternative medicine by asthma patients. QJM. 2003 Oct;96(10):747-54. doi: 10.1093/qjmed/hcg121. PMID 14500861
- [Background] Jonas WB, Kaptchuk TJ, Linde K. A critical overview of homeopathy. Ann Intern Med. 2003 Mar 4;138(5):393-9. doi: 10.7326/0003-4819-138-5-200303040-00009. PMID 12614092
- [Background] McCarney RW, Linde K, Lasserson TJ. Homeopathy for chronic asthma. Cochrane Database Syst Rev. 2004;2004(1):CD000353. doi: 10.1002/14651858.CD000353.pub2. PMID 14973954
- [Background] Ernst E. Is reflexology an effective intervention? A systematic review of randomised controlled trials. Med J Aust. 2009 Sep 7;191(5):263-6. doi: 10.5694/j.1326-5377.2009.tb02780.x. PMID 19740047
- [Background] Brygge T, Heinig JH, Collins P, Ronborg S, Gehrchen PM, Hilden J, Heegaard S, Poulsen LK. Reflexology and bronchial asthma. Respir Med. 2001 Mar;95(3):173-9. doi: 10.1053/rmed.2000.0975. PMID 11266233
- [Background] Lewith GT, Watkins AD, Hyland ME, Shaw S, Broomfield JA, Dolan G, Holgate ST. Use of ultramolecular potencies of allergen to treat asthmatic people allergic to house dust mite: double blind randomised controlled clinical trial. BMJ. 2002 Mar 2;324(7336):520. doi: 10.1136/bmj.324.7336.520. PMID 11872551
- [Background] White A, Slade P, Hunt C, Hart A, Ernst E. Individualised homeopathy as an adjunct in the treatment of childhood asthma: a randomised placebo controlled trial. Thorax. 2003 Apr;58(4):317-21. doi: 10.1136/thorax.58.4.317. PMID 12668794